CLINICAL TRIAL: NCT01559207
Title: Reproducibility of Plasma Nucleosomes and Free DNA as Markers for Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2011/SB-02; 2012-A00198-35 (Other: ANSM)
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Venous Thromboembolism
Keywords: nucleosome; plasma nucleosome concentrations; free DNA; plasma free DNA concentrations
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA, CTAD and dry tubes; Biological collection at the Nîmes University Hospital.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with VTE: Group "P" is composed of all patients with a history of VTE. Group "Px" is a subgroup of 15 patients from group P. Members of "Px" are randomly selected from "P".
- Healthy volunteers: Group "T": 15 healthy volunteers with no history of VTE will be included in this group.

SUMMARY:
The main objective of this study is to evaluate, for 15 healthy volunteers and for 15 patients with a history of venous thromboembolism (VTE), the monthly variation (over 6 months) of plasma nucleosome and free DNA concentrations.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To describe, for 15 healthy volunteers with no history of venous thromboembolism (VTE), plasma nucleosome and DNA concentrations.

B. To describe, for 100 patients with a history of VTE currently consulting for chronic disease or thrombophilia work-up, plasma nucleosome and DNA concentrations.

C. To compare plasma nucleosome and DNA concentrations between healthy volunteers and VTE patients

D. To describe, for 100 patients with a history of VTE currently consulting for chronic disease or thrombophilia work-up, the relationships between classification of VTE and plasma nucleosome concentrations:

* anatomical classification of VTE: (i)superficial, deep ((ii)distal or (iii)proximal), or (iv)pulmonary embolism
* circumstantial classification of VTE: (i) triggered, no chronic risk factor; (ii) untriggered, with chronic risk factor; (iii)triggered, with chronic risk factor; (iv) untriggered, no chronic risk factor (idiopathic)

E. To describe, for 100 patients with a history of VTE, the variation in plasma nucleosome concentrations 6 months after the first evaluation

* according to the above anatomical classification
* according to the above circumstantial classification
* according to intercurrent events and treatments

F. To compare the plasma concentrations of nucleosomes and free DNA

G. To evaluate the relationship between plasma nucleosome and free DNA concentrations and:

* circulating leukocyte populations: total leukocyte count, absolute number of neutrophils, monocytes, lymphocytes
* markers of coagulation activation: d-dimers, circulating fibrin monomers
* platelet count
* patients on antivitamin K: INR, patients receiving heparin: antiXa activity

H. Creation of a biological collection

ELIGIBILITY:
Inclusion Criteria:

* The patient or volunteer must have given his/her informed and signed consent
* The patient or volunteer must be insured or beneficiary of a health insurance plan
* The patient or volunteer is available for 6 months of follow-up

For group "P":

* patient with a history of VTE

For group "T":

* healthy volunteer
* no history of VTE
* no history of chronic disease
* no history of neoplastic disease
* no history of chronic infection
* not taking anticoagulants, antiplatelet medications
* no acute disease or infection during the last 2 weeks

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient gave birth in the past three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is composed of 15 healthy volunteers with no history of VTE (group "T") and 100 patients with VTE (group "P"). Fifteen randomly selected members of group P make up the sub-group "Px".
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10-20 (Actual); Study Completion 2014-10-20 (Actual)

PRIMARY OUTCOMES:
Plasma nucleosome concentration (ng/ml) | baseline
  For cohortes T and P
Plasma nucleosome concentration (ng/ml) | 6 months
  For cohortes T and P
Plasma nucleosome concentration (ng/ml) | 1 month
  For cohortes T and Px
Plasma nucleosome concentration (ng/ml) | 2 months
  For cohortes T and Px
Plasma nucleosome concentration (ng/ml) | 3 months
  For cohortes T and Px
Plasma nucleosome concentration (ng/ml) | 4 months
  For cohortes T and Px
Plasma nucleosome concentration (ng/ml) | 5 months
  For cohortes T and Px
Plasma free DNA concentration (ng/ml) | baseline
  For cohortes T and P
Plasma free DNA concentration (ng/ml) | 6 months
  For cohortes T and P
Plasma free DNA concentration (ng/ml) | 1 month
  For cohortes T and Px
Plasma free DNA concentration (ng/ml) | 2 months
  For cohortes T and Px
Plasma free DNA concentration (ng/ml) | 3 months
  For cohortes T and Px
Plasma free DNA concentration (ng/ml) | 4 months
  For cohortes T and Px
Plasma free DNA concentration (ng/ml) | 5 months
  For cohortes T and Px

SECONDARY OUTCOMES:
Hemogram | baseline
  hemoglobin, platelet count, leukocytes, polynuclear neutrophils, mean corpuscular volume, monocytes, mean corpuscular hemoglobin, lymphocytes, polynuclear eosinophils, polynuclear basophils
Hemogram | 6 months
  hemoglobin, platelet count, leukocytes, polynuclear neutrophils, mean corpuscular volume, monocytes, mean corpuscular hemoglobin, lymphocytes, polynuclear eosinophils, polynuclear basophils
Hemogram | 1 month
  hemoglobin, platelet count, leukocytes, polynuclear neutrophils, mean corpuscular volume, monocytes, mean corpuscular hemoglobin, lymphocytes, polynuclear eosinophils, polynuclear basophils
Hemogram | 2 months
  for cohortes "T" and "Px": hemoglobin, platelet count, leukocytes, polynuclear neutrophils, mean corpuscular volume, monocytes, mean corpuscular hemoglobin, lymphocytes, polynuclear eosinophils, polynuclear basophils
Hemogram | 3 months
  for cohortes "T" and "Px": hemoglobin, platelet count, leukocytes, polynuclear neutrophils, mean corpuscular volume, monocytes, mean corpuscular hemoglobin, lymphocytes, polynuclear eosinophils, polynuclear basophils
Hemogram | 4 months
  for cohortes "T" and "Px": hemoglobin, platelet count, leukocytes, polynuclear neutrophils, mean corpuscular volume, monocytes, mean corpuscular hemoglobin, lymphocytes, polynuclear eosinophils, polynuclear basophils
Hemogram | 5 months
  for cohortes "T" and "Px": hemoglobin, platelet count, leukocytes, polynuclear neutrophils, mean corpuscular volume, monocytes, mean corpuscular hemoglobin, lymphocytes, polynuclear eosinophils, polynuclear basophils
D-dimers (ng/ml) | baseline
D-dimers (ng/ml) | 6 months
D-dimers (ng/ml) | 1 months
  cohortes "T" and "Px" only
D-dimers (ng/ml) | 2 months
  cohortes "T" and "Px" only
D-dimers (ng/ml) | 3 months
  cohortes "T" and "Px" only
D-dimers (ng/ml) | 4 months
  cohortes "T" and "Px" only
D-dimers (ng/ml) | 5 months
  cohortes "T" and "Px" only
Fibrin monomers (ng/ml) | baseline
Fibrin monomers (ng/ml) | 6 months
Fibrin monomers (ng/ml) | 1 month
  cohortes "T" and "Px" only
Fibrin monomers (ng/ml) | 2 months
  cohortes "T" and "Px" only
Fibrin monomers (ng/ml) | 3 months
  cohortes "T" and "Px" only
Fibrin monomers (ng/ml) | 4 months
  cohortes "T" and "Px" only
Fibrin monomers (ng/ml) | 5 months
  cohortes "T" and "Px" only
creatininemia (µM/L) | baseline
creatininemia (µM/L) | 6 months
blood Glutamo-oxaloacetate transaminase (UI/L) | baseline
blood Glutamo-oxaloacetate transaminase (UI/L) | 6 months
blood glutamo-pyruvate transaminase (UI/L) | baseline
blood glutamo-pyruvate transaminase (UI/L) | 6 months
blood gamma-glutamyl transaminase (UI/L) | 6 months
blood gamma-glutamyl transaminase (UI/L) | baseline
C reactive protein (mg/l) | baseline
C reactive protein (mg/l) | 6 months
blood fibrinogen (g/l) | baseline
blood fibrinogen (g/l) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Bouvier, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Bouvier S, Bastide S, Chouirfa S, Nouvellon E, Mercier E, Bigot L, Lavigne G, Cayla G, Perez-Martin A, Gris JC. Reliability of hemostasis biomarkers is affected by time-dependent intra-patient variability. J Thromb Haemost. 2018 Jun 8. doi: 10.1111/jth.14198. Online ahead of print. PMID 29883046